CLINICAL TRIAL: NCT05424952
Title: The Effectiveness of Conversational AI Service (chatbot) Utilization on Vaccine Confidence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: National University of Singapore (Other); Health Intervention and Technology Assessment Program (HITAP) (Unknown)
Responsible Party: Principal Investigator, Joseph Tsz Kei Wu, Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: UW 21-659
Record Dates: First submitted 2021-12-21; First posted 2022-06-21 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Vaccination Hesitancy
MeSH Terms: conditions — Vaccination Hesitancy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (No Intervention): Eligible adults with unvaccinated senior parents/grandparents or children.
- Intervention (Experimental): Eligible adults with unvaccinated senior parents/grandparents or children.
  Interventions: Other: Conversational AI Service (Chatbot)

INTERVENTIONS:
Other: Conversational AI Service (Chatbot) — WhatsApp or Messenger Chatbot for COVID-19 vaccines
  Arms: Intervention

SUMMARY:
The primary objective of this study is to develop and evaluate a conversational AI service (chatbot) on social media platforms to obtain accurate and up-to-date vaccine information, and assess the impact of chatbot usage on users' vaccine confidence and acceptance in Hong Kong, Singapore, and Thailand.

DETAILED DESCRIPTION:
The investigators will focus on vulnerable seniors and/or children from Hong Kong, Singapore and Thailand who have refused or delayed COVID-19 vaccination. Participants will be recruited by an online panel to meet the target quota by age and sex. Participants will then be randomly assigned to the intervention group and the control group. For both intervention and control groups, evaluation questionnaires will be given out to the study participants asking questions about their demographics, including age, sex, educational level, employment status and household income levels. Participants will then answer questions regarding COVID-19 vaccine confidence, including the effectiveness and safety of vaccines, and the motivations of the policymakers who decided on the needed vaccines. Participants will be asked about COVID-19 vaccine acceptance including the intention to receive COVID-19 vaccines, make plans to receive COVID-19 vaccines, and receive at least one dose of COVID-19 vaccines. The intervention group will then be asked to use the chatbot developed by the research team for up to two weeks. The chatbot is developed under the RE-AIM framework for formative, impact, and process evaluation of the intervention. The control group will have no exposure to the chatbot.

The chatbot will be supported with data from 1) social listening analytics for monitoring local real-time discourses in the digital space on COVID-19 vaccine hesitancy and misinformation, and 2) formative, baseline, and endpoint evaluation, which will generate evidence for development and improvement/refinement.

ELIGIBILITY:
Inclusion Criteria:

* Hong Kong adult residents (English or Chinese users) with (a) unvaccinated senior parents/grandparents aged 60 (including those who received first dose after the announcement of the COVID passport on 4th of January) or (b) unvaccinated children aged below 18.
* Thailand adult residents (Thai users) with (a) unvaccinated senior parents/grandparents aged 60 or above or (b) unvaccinated children aged below 18.
* Singapore adult residents (English or Chinese users) with unvaccinated children aged between 5 to 11 years old.

Exclusion Criteria:

* People who do not meet the inclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1000 (Actual)
Dates: Start 2022-02-11 (Actual); Primary Completion 2023-02-17 (Actual); Study Completion 2023-02-17 (Actual)

PRIMARY OUTCOMES:
Covid-19 vaccines confidence Index | 1 week
  1. "Overall, I think COVID-19 vaccines are important for children/senior parents (or grandparents)"
  2. "Overall, I think COVID-19 vaccines are safe for children/parents (or grandparents)"
  3. "Overall, I think COVID-19 vaccines are effective for children/parents (or grandparents)"
  The response is a 5-point Likert scale: (a) Strongly agree (b)Tend to agree (c) Do not know (d) Tend to disagree (e) Strongly disagree
Covid-19 vaccines acceptance | 1 week
  1. What is the vaccination status of your children/senior parents (or grandparents) as of now?
     1. Is vaccinated with at least the first dose of the vaccine
     2. Has made an appointment but has not been vaccinated with the first dose yet
     3. Has not made an appointment but will get the vaccine.
     4. Has no plan to get vaccinated anytime soon.
  2. Do you want your children/senior parents (or grandparents) vaccinated against COVID-19 if vaccination is indicated and available for them?
     1. Yes, definitely.
     2. Unsure, but leaning towards yes.
     3. Unsure, but leaning towards no.
     4. No, definitely not.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph T Wu, PhD, Principal Investigator — The University of Hong Kong
Locations (3):
- The University of Hong Kong, Hong Kong, Hong Kong
- National University of Singapore, Singapore, Singapore
- Health Intervention and Technology Assessment Program, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in the article, after de-identification (text, tables, figures, and appendices), will be shared. A written data-sharing request for meta-analysis should be submitted by email with a methodologically sound proposal. Proposals should be directed to kathysleung@connect.hku.hk; to gain access, data requestors will need to sign a data access agreement.
Supporting Information: Study Protocol
Time Frame: Beginning 9 months and ending 36 months following article publication
Access Criteria: Researchers who provide a methodologically sound proposal for meta-analysis. Proposals should be directed to Kathyleung@connect.hku.hk; to gain access, data requestors will need to sign a data access agreement.

REFERENCES:
- [Background] Glasgow RE, Vogt TM, Boles SM. Evaluating the public health impact of health promotion interventions: the RE-AIM framework. Am J Public Health. 1999 Sep;89(9):1322-7. doi: 10.2105/ajph.89.9.1322. PMID 10474547
- [Background] Gaglio B, Shoup JA, Glasgow RE. The RE-AIM framework: a systematic review of use over time. Am J Public Health. 2013 Jun;103(6):e38-46. doi: 10.2105/AJPH.2013.301299. Epub 2013 Apr 18. PMID 23597377
- [Background] Kobayashi T, Nishina Y, Tomoi H, et al. Corowa-kun: Impact of a COVID-19 vaccine information chatbot on vaccine hesitancy, Japan 2021. medRxiv 2021: 2021.05.26.21257854.
- [Background] de Figueiredo A, Simas C, Karafillakis E, Paterson P, Larson HJ. Mapping global trends in vaccine confidence and investigating barriers to vaccine uptake: a large-scale retrospective temporal modelling study. Lancet. 2020 Sep 26;396(10255):898-908. doi: 10.1016/S0140-6736(20)31558-0. Epub 2020 Sep 10. PMID 32919524
- [Background] Larson HJ, Smith DM, Paterson P, Cumming M, Eckersberger E, Freifeld CC, Ghinai I, Jarrett C, Paushter L, Brownstein JS, Madoff LC. Measuring vaccine confidence: analysis of data obtained by a media surveillance system used to analyse public concerns about vaccines. Lancet Infect Dis. 2013 Jul;13(7):606-613. doi: 10.1016/S1473-3099(13)70108-7. Epub 2013 May 13. PMID 23676442
- [Background] Wang Q, Yang L, Jin H, Lin L. Vaccination against COVID-19: A systematic review and meta-analysis of acceptability and its predictors. Prev Med. 2021 Sep;150:106694. doi: 10.1016/j.ypmed.2021.106694. Epub 2021 Jun 22. PMID 34171345
- [Background] Zhang J, Featherstone JD, Calabrese C, Wojcieszak M. Effects of fact-checking social media vaccine misinformation on attitudes toward vaccines. Prev Med. 2021 Apr;145:106408. doi: 10.1016/j.ypmed.2020.106408. Epub 2021 Jan 1. PMID 33388335
- [Background] Altay S, Hacquin AS, Chevallier C, Mercier H. Information delivered by a chatbot has a positive impact on COVID-19 vaccines attitudes and intentions. J Exp Psychol Appl. 2023 Mar;29(1):52-62. doi: 10.1037/xap0000400. Epub 2021 Oct 28. PMID 34726454
- [Background] Thomala LL. Penetration rate of leading social networks in Hong Kong as of 3rd quarter 2020 (Link: https://www.statista.com/statistics/412500/hk-social-network-penetration/, last accessed on August 1, 2021). Statista; 2020.
- [Background] Kemp S. Digital 2021: Hong Kong (Link: https://datareportal.com/reports/digital-2021-hong-kong, last accessed on August 1, 2021). Data Reportal; 2021.
- [Background] Müller J. Social network penetration in Singapore Q3 2020 (Link: https://www.statista.com/statistics/284466/singapore-social-network-penetration/, last accessed on August 1, 2021). Statista; 2020.
- [Background] Huang C. Hong Kong faces uphill task to vaccinate its seniors against Covid-19 (Link: https://www.straitstimes.com/asia/east-asia/hong-kongs-uphill-push-to-vaccinate-its-seniors-against-covid-19, last accessed on August 1, 2021). The Straits Times. 2021.
- [Background] Steve. Lexicon. The LINE Phenomenon in Thailand - By the Numbers (Link: https://lexiconthai.com/blog/the-line-phenomenon-in-thailand-by-the-numbers/, last accessed on August 1, 2021), 2020.
- [Background] Agency T. Line in Thailand Internet Population (Link: https://www.twfdigital.com/blog/2020/04/line-user- stat-in-thailand-2020/, last accessed on August 1, 2021), 2020.
- [Background] Get bad news (Link: https://www.getbadnews.com/#intro, last accessed on August 1, 2021). 2021.
- [Background] Elkin J. WHO launches a chatbot on Facebook Messenger to combat COVID-19 misinformation. (Link: https://www.who.int/news-room/feature-stories/detail/who-launches-a-chatbot-powered-facebook- messenger-to-combat-covid-19-misinformation, last accessed: August 1, 2021). 2020.
- [Background] Larson HJ, Schulz WS, Tucker JD, Smith DM. Measuring vaccine confidence: introducing a global vaccine confidence index. PLoS Curr. 2015 Feb 25;7:ecurrents.outbreaks.ce0f6177bc97332602a8e3fe7d7f7cc4. doi: 10.1371/currents.outbreaks.ce0f6177bc97332602a8e3fe7d7f7cc4. PMID 25789200
- [Background] SAGE. Report of the SAGE Working Group on Vaccine Hesitancy (Link: https://www.who.int/immunization/sage/meetings/2014/october/1_Report_WORKING_GROUP_vaccine_hesita ncy_final.pdf, last accessed on August 1, 2021), 2014.